CLINICAL TRIAL: NCT01776996
Title: An Expanded Access Protocol for Subjects Who Have Completed Clinical Studies Involving Maraviroc
Status: No longer available | Type: Expanded Access
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116278
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Expanded access, HIV, maraviroc
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Continued Access Arm — All subjects will be on maraviroc 300 mg twice a day, unless a dose adjustment is required due to certain concomitant medications. For those subjects in South Africa and Argentina who were previously receiving Combivir along with maraviroc in Study A4001026, Combivir will be supplied as tablets containing 150 mg lamivudine and 300 mg zidovudine. One Combivir tablet will be taken orally twice a day.

SUMMARY:
This is an open-label protocol designed to provide continued access to maraviroc to only those subjects who have completed previous studies of maraviroc and continue to receive clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Subject has participated in a clinical trial that evaluated maraviroc and is continuing to derive clinical benefit from maraviroc treatment.
* Subject must agree to use an acceptable method of contraception for the duration of the study as outlined at the end of the inclusion criteria.
* Subject agrees to the specified study procedures.

Exclusion Criteria:

* Subject who is an investigational site staff member or an employee of the Sponsor that is directly involved in the conduct of the trial.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Contra-indications to use of maraviroc as described in the Investigator Brochure.
* Past documented dual/mixed or C-X-C chemokine receptor type 4 HIV tropism.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (25):
- Argentina (3):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Modena
- GSK Investigational Site, Bydgoszcz, Poland
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, N.Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
- South Africa (9):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Gauteng, Gauteng
  - GSK Investigational Site, Soweto, Gauteng
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Port Elizabeth
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Pretoria North
  - GSK Investigational Site, Westdene
- Switzerland (3):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Lugano
  - GSK Investigational Site, Zurich